CLINICAL TRIAL: NCT03731078
Title: Pilot Study of Cognitive Behavioral Therapy-Informed Physical Therapy Intervention in Functional Neurological Disorders
Status: Terminated | Type: Observational
Why Stopped: Study as designed did not prove feasible with the challenges faced amidst the COVID-19 pandemic
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Lewis Perez, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2018P001674
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Functional Neurological Disorder
Keywords: Conversion Disorder; Functional Limb Weakness; Functional Movement Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Motor Functional Neurological Disorder: The cohort will consist of patients with clinically-established motor functional neurological disorder, which includes individuals with functional movement disorders and functional limb weakness. Individuals with functional movement disorders and/or functional limb weakness who also have psychogenic nonepileptic seizures will be included. Patients will receive CBT informed PT intervention. The physical therapy intervention will be usual care in FND and based on consensus recommendations, clinical trials and good practices.
  Interventions: Other: CBT Informed physical therapy Intervention

INTERVENTIONS:
Other: CBT Informed physical therapy Intervention — The 12 physical therapy sessions delivered in Massachusetts General Hospital outpatient physical therapy sites sessions include:1) evaluation and education; 2) strategy identification and goal setting; 3) functional strengthening part one; 4) functional strengthening part two; 5) pre-gait activities with distraction; 6) gait training with distraction and use of strategies; 7) minimizing tremor with use of strategies; 8) higher level balance training; 9) functional reintegration part one; 10) functional reintegration part two; 11) identification of strategies to limit recurrence; 12) education for relapse prevention.Patients will also be given and asked to complete the self-guided CBT workbookL Overcoming Functional Neurological Symptoms: A Five Area Approach. They will be asked to complete the first two chapters over the first 4 weeks and the remaining 8 chapters over the following 8 weeks.

SUMMARY:
Functional Neurological Disorder (FND/ Conversion Disorder) is a highly prevalent and disabling neuropsychiatric condition. Motor FND symptoms include Functional Movement Disorders (FMD) and Functional Weakness and Psychogenic Nonepileptic Seizures (PNES).Though patients with FND present with a wide variety of symptoms, FMD, PNES, and functional weakness may be viewed as overlapping conditions lying along a phenotypic spectrum for a single disorder. Patients with FND frequently present with psychiatric symptoms, including depression, anxiety, Borderline Personality Disorder, and Post-Traumatic Stress Disorder, alongside their physical symptoms. To treat these symptoms, patients with FND are frequently enrolled in physical therapy and cognitive behavioral therapy, which are considered usual care for FND at our center. Developing a further understanding of treatment outcome, including biomarkers of clinical improvement and psychometric factors associated with treatment response, could inform future interventions and better tailor treatments to patients with specific FND symptom profiles.

We hypothesize that treatment response will be associated with structural and functional alterations in salience network regions and that more adaptive neuropsychiatric profiles at baseline will predict a positive treatment outcome.

DETAILED DESCRIPTION:
Functional Neurological Disorder (FND) (Conversion Disorder) is a poorly understood and prevalent somatoform disorder, making up 16% of outpatient neurology referrals. Patients with motor FND (mFND) are difficult to treat, result in major morbidity, and are costly to the US. An estimated $256 billion is spent annually treating this population. mFND includes Functional Movement Disorders (FMD), Functional Weakness (FW) and Psychogenic Nonepileptic Seizures (PNES).

This project will investigate brain network profiles associated with and predictive of clinical improvement in patients with Functional Neurological Disorder (FND) following a 12-week cognitive behavioral therapy-informed physical therapy treatment program. Integrated physical therapy along with self-guided cognitive behavioral therapy is usual care for patients with FND experiencing motor symptoms at the Massachusetts General Hospital. Patients with motor FND experience significant impairment and often face issues with treatment management. Recent advancements in clinical research, catalyzed by new diagnostic criteria and an updated care model, have emphasized physical therapy and cognitive behavioral therapy as important evidence-based treatments for this population. Additionally, developments in neuroscience have allowed for a more comprehensive understanding of the neurobiology of FND. However, there has been limited investigation of longitudinal biomarkers associated with and predictive of treatment response, highlighting the need for an improved understanding of neurobiological changes underlying prognosis in FND.

We propose acquiring structural and functional brain imaging data in combination with psychometric assessments and patient chart review to examine neurobiological mechanisms of associated with participation in a cognitive behavioral therapy-informed physical therapy treatment program for patients with FND.

Primary Aim and Hypotheses The primary goal of this study is to provide structural and functional biomarkers related to and predictive of treatment response and clinical outcome in patients with motor FND following a 12-week cognitive behavioral therapy-informed physical therapy treatment program (usual care).

Specific Aim 1:

SA1) Identify structural MRI biomarkers linked to and predictive of improvement following cognitive behavioral therapy-informed physical therapy in FND.

Hypotheses: Improvement will correlate with increased volume, cortical thickness, and/or white matter integrity in salience network-related regions post- versus pre- treatment. Pre-treatment (baseline) salience network volume, cortical thickness, and/or white mater integrity will predict clinical outcome of the 12-week treatment program.

Specific Aim 2:

SA2) Identify resting-state functional MRI biomarkers linked to and predictive of improvement following cognitive behavioral therapy-informed physical therapy in FND.

Hypotheses: Improvement will correlate with reduced post- versus pre- treatment salience-somatomotor network resting state functional connectivity, and pre-treatment salience-somatomotor network functional connectivity strength will predict clinical outcome.

SA3) Identify baseline psychometric factors that correlate with clinical improvement (post vs. pre-treatment), including differences among FND sub-populations and baseline predictors of clinical improvement in FND.

Hypotheses: FND patients with more adaptive psychological profiles at baseline will be more responsive to treatment.

ELIGIBILITY:
Inclusion Criteria:

* FND patients will be recruited from the FND clinic and allied neurology and psychiatry clinics at Massachusetts General Hospital, with additional recruitment occurring through the physical therapy department. This study aims to recruit a total of 70 patients with motor FND. FND subjects will meet established clinical diagnostic criteria and patients with functional weakness will be diagnosed by "positive" signs suggestive of functional weakness including but not limited to a positive Hoover's sign. Individuals with PNES who have a concurrent functional limb weakness and/or a functional movement disorder will also be recruited. In addition, all individuals will have a clinical indication for PT (i.e. limb weakness, gait difficulties, abnormal movements).

Exclusion Criteria:

* Any significant major neurological disorder resulting in specific MRI abnormalities (i.e. encephalomalacia, severe traumatic brain injury (TBI)), poorly controlled major medical illness with known central nervous system consequences, inability to read English, pregnancy, claustrophobia, or inability to satisfy MRI safety measures. Additionally, patients with isolated PNES will not be considered for this study.

Note: individuals who are eligible for the study but have an MRI contraindication may be offered study enrollment with MRI data collection for participation in aim 3 of this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: motor functional neurological disorder
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Short Form Health Survery 36 (SF-36) | 1-5 years
  questionnaire to identify change in health-related quality of life post vs. pre-treatment

SECONDARY OUTCOMES:
Screening for Somatoform Symptoms Conversion Disorder subscale (SOMS:CD) | 1-5 years
  composite score post vs. pre-treatment
Patient Health Questionnaire-15 (PHQ-15) | 1-5 years
  composite score post vs. pre-treatment
Clinical Global Impressions (CGI) - clinician rated scale | 1-5 years
  clinical global impression of improvement as rated by clinician
Clinical Global Impressions (CGI) - patient rated | 1-5 years
  clinical global impression of improvement as rated by patient
10meter walk test | 1-5 years
  change in post vs. pre-treatment speed of walking at preferred pace
Five Times Sit to Stand test | 1-5 years
  change in post vs. pre-treatment time to move from sitting to standing five times
Simplified Functional Movement Disorders Rating Scale (S-FMDRS) | 1-5 years
  clinician rated functional neurological symptom severity scale

CONTACTS AND LOCATIONS:
Overall Officials: David L Perez, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No